CLINICAL TRIAL: NCT01534676
Title: Harmful Effects of Transfusion of Older Stored Red Cells: Iron and Inflammation
Brief Title: Effects of Transfusion of Older Stored Red Cells
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting donors and recipients, looking for alternative sites
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Steven L. Spitalnik, Professor of Pathology and Cell Biology, Columbia University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAI1111; R01HL098014 (NIH)
Record Dates: First submitted 2012-02-14; First posted 2012-02-17 (Estimated); Results first posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-08

CONDITIONS: Sickle Cell Disease; Thalassemia
Keywords: iron; transfusion; red blood cells; sickle cell disease; thalassemia; blood donors
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia | interventions — Blood Transfusion; Blood Specimen Collection; Chelation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Transfusion of Fresh blood (Active Comparator): The recipient will receive one or two units of fresh blood <14 days old, as per their chronic transfusion schedule - on or off chelation therapy.
  Interventions: Procedure: Transfusion; Biological: Blood; Procedure: Chelation therapy
- Transfusion of Stored blood (Experimental): The recipient will receive one or two units of old blood >28 days old, as per their chronic transfusion schedule - on or off chelation therapy.
  Interventions: Procedure: Transfusion; Biological: Blood; Procedure: Chelation therapy
- Transfusion of Cryopreserved Blood (Active Comparator): The recipient will receive one or two units of cryopreserved (fresh/old) blood, as per their chronic transfusion schedule - off chelation therapy.
  Interventions: Procedure: Transfusion; Biological: Blood
- Transfusion of Washed Blood (Active Comparator): The recipient will receive one or two units of washed (fresh/old) stored blood >28 days old, as per their chronic transfusion schedule - off chelation therapy.
  Interventions: Procedure: Transfusion; Biological: Blood

INTERVENTIONS:
Procedure: Transfusion — A routine medical procedure to transfuse packed red blood cells.
  Other Names: RBC transfusion
Biological: Blood — Processing of RBC for transfusion include the following:
  * Fresh
  * Stored
  * Washed
  * Frozen (Cryopreserved)
  Other Names: RBC product; Reb Blood Cells
Procedure: Chelation therapy — (non-experimental) A medical procedure that involves the administration of chelating agents to remove heavy metals from the body.
  Arms: Transfusion of Fresh blood; Transfusion of Stored blood

SUMMARY:
The purpose of this study is to determine the effects of transfusion of fresh and stored blood on patients.

The investigators hope to test:

* whether a similar effect (older stored blood is associated with worse outcomes) is seen in chronically transfused patients with hemoglobinopathies. This patient population will also allow the investigators to test whether iron- chelation therapy is beneficial in this setting.
* whether washing or cryopreserving the red blood cells has any effect on this outcome.

These findings may explain the immunomodulatory effects of older stored blood in patients and will help us develop safer transfusion products for patients.

DETAILED DESCRIPTION:
Epidemiologic studies suggest that older stored blood is associated with worse outcomes in certain hospitalized patients. Storage of red cells is associated with a storage lesion and the survival of transfused red cells decreases with increasing storage time, thus older blood is associated with an increased acute delivery of hemoglobin-iron to the reticuloendothelial system. The investigators have preliminary data in healthy human volunteers suggesting that delivery of a significant iron load to the reticuloendothelial system from aged red cells leads to the elaboration of a potentially toxic form of iron known as non-transferrin-bound iron.

ELIGIBILITY:
Inclusion Criteria (Recipient):

* specific, well-characterized hemoglobinopathy
* chronic simple transfusion therapy (transfusion episodes < 6 weeks apart in frequency)
* chronic iron chelation therapy
* not pregnant by self-report and not planning pregnancy
* age > 1 year old

Exclusion Criteria (Recipient):

* clinically unstable
* treatment for mental illness
* imprisonment
* institutionalization

Inclusion Criteria (Donor):

* 21-65 years of age
* male weight > 130 lbs, female weight > 150 lbs
* male height > 5'1", female height > 5'5"
* hemoglobin > 15.0 g/dL
* reasonably certain of intention to stay in New York City metropolitan area for study duration
* previously tolerated red blood cell donation

Exclusion Criteria (Donor):

* ineligible for donation based on New York Blood Center blood donor screening questionnaire
* systolic blood pressure < 90 or > 180 mm Hg, diastolic blood pressure < 50 or > 100 mm Hg
* heart rate < 50 or > 100
* temperature > 99.5 F prior to donation
* positive by standard infectious disease testing performed on blood donors

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Spitalnik, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a research study carried out at Columbia University Medical Center. Participants with a blood disorder and currently receive blood transfusions as treatment will be transfused fresh, stored, washed or frozen blood according to regular schedule for up to 3 years. Volunteer dedicated donors will also be asked to provide consent.
Pre-assignment Details: Enrolled participants (recipients) were never randomized or received transfusion on study because study closed due to poor enrollment.
Groups:
- Recipients: Participants with a blood disorder (either sickle cell disease or thalassemia) and currently receive blood transfusions as treatment - will be receiving the following transfusion according to regular schedule: a fresh blood, a stored blood, a washed blood, and a frozen blood transfusion.
- Donors: Volunteer dedicated donors will be recruited to donate blood for each transfusion events over the next 3 years. Each patient with a chronic illness such as sickle cell disease or thalassemia will have one dedicated donor.
Period: Overall Study
Arm/Group | Recipients | Donors
Started | 2 | 1
Completed | 0 | 0
Not Completed | 2 | 1
Not completed — Study closed due to poor enrollment | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Recipients | Donors | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 2
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Non-transferrin-bound Iron Level
Time Frame: 2 hours after transfusion
Population: Enrolled participants (recipients) were never randomized or received transfusion on study because study closed due to poor enrollment. No data was collected or analyzed.
Arm/Group | Recipients | Donors
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Recipients | Donors
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes